CLINICAL TRIAL: NCT01984385
Title: Hip Fracture Impact on Vascular Events In Noncardiac Surgery patIents: a cOhort evaluatioN (Hip VISION): Pilot Study
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, P.J. Devereaux, MD, PhD, FRCP(C), Population Health Research Institute
Other Study IDs: HipVISION Pilot - 2013
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a hip fracture

SUMMARY:
Hip VISION (Pilot Study) is a Prospective Observational Cohort Study to evaluate the incidence of overall and cause-specific mortality among consecutive patients aged ≥ 18 years presenting with hip fracture to the Juravinski Hospital of the Hamilton Health Sciences. This pilot study will assess the feasibility of a larger prospective international cohort study. After eligibility has been confirmed and informed consent has been obtained, participants will be registered in the study. Troponin level, complete blood counts and serum creatinine level will be collected at day 1 through day 10 post admission. CAM instrument will be employed at admission and once daily post admission day 1 through day 10. FIM Instrument will be administered within 72 hours of admission to establish pre-fracture functional independence and disability. Patients will be contacted by research personnel by telephone 30 days after study registration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years with hip fractures (i.e. fractures involving the subcapital, femoral neck, or intertrochanteric regions), treated either operatively or non-operatively
2. Mechanism of injury consistent with either:

   1. A fall from a standing height or;
   2. Another mechanism of injury which, in the clinical judgment of an orthopedic surgeon, would impart the same or less traumatic energy as a fall from a standing height

Exclusion Criteria:

1. Patients with fractures isolated to the proximal femoral shaft, with no involvement of the intertrochanteric, femoral neck, or subcapital region
2. Patients with hip fractures resulting from high energy mechanisms, such as motor vehicle accidents or falls from a substantial height
3. Patient who refuse 30-day or 6-month follow up
4. Patients who refuse to consent either by themselves or through a substitute decision-maker (for patients unable to consent, we will use a deferred consent process, as described below).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total and cause specific mortality in hip fracture patients at 30 days | 30 days
Major complications within 30 days. | 30 days
  Composite of vascular mortality, nonfatal MI, nonfatal stroke, nonfatal PE, sepsis, and life-threatening bleeding.

SECONDARY OUTCOMES:
Nonfatal myocardial infarction | 30 days
Nonfatal myocardial injury after noncardiac surgery | 30 days
Nonfatal pulmonary embolism | 30 days
Nonfatal infection | 30 days
Nonfatal bleeding | 30 days
Nonfatal stroke | 30 days
New congestive heart failure | 30 days
New atrial fibrillation | 30 days
Nonfatal cardiac arrest | 30 days
Deep vein thrombosis | 30 days
New acute renal failure requiring dialysis | 30 days
Cardiac catheterization | 30 days
PCI | 30 days
CABG | 30 days
CAM days 1-7 post-op | 1-7 days post-op
Implant failure or periprosthetic fracture | 30 days
Re-operation | 30 days
Length of hospital stay | 30 days
New nursing home residence | 30 days
First mobilization | 30 days
FIM (motor function) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: PJ Devereaux, PhD, Principal Investigator — Population Health Research Institute
Locations (1):
- Juravinski Hospital and Cancer Centre (HHS), Hamilton, Ontario, Canada